CLINICAL TRIAL: NCT06927544
Title: A Randomised Clinical Trial of Surgical Methods and Intraocular Gas Tamponade for Treatment of Large (410-1000 μm) Idiopathic Macular Holes
Brief Title: Intraocular Gas Tamponade for Treatment of Large Idiopathic Macular Holes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Filatov Institute of Eye Diseases and Tissue Therapy (Other)
Collaborators: Ukrainian Vitreoretinal Society (Other)
Responsible Party: Principal Investigator, Mykola Umanets, Mykola Umanets, MD, PhD, Head of Department of Retina and Vitreous Pathology SI "The Filatov Institute of Eye Diseases and Tissue Therapy", President of Ukrainian Vitreoretinal Society, The Filatov Institute of Eye Diseases and Tissue Therapy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23/12/2024
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Macular Hole; Macular Hole; Macular Holes; Full Thickness Macular Hole
Keywords: macular hole; pars plana vitrectomy; perfluoropropane (C3F8); sulfur hexafluoride (SF6); Idiopathic Macular Hole; Full thickness macular hole; large macular hole; large macular holes
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perfluoropropane (15% C3F8) gas tamponade (Other): Macular hole surgery with ILM-peeling and 15% C3F8 gas tamponade
  Interventions: Procedure: Pars plana vitrectomy
- Hexafluoride (20% SF6) gas tamponade (Other): Macular hole surgery with ILM-peeling and hexafluoride (20% SF6) gas tamponade
  Interventions: Procedure: Pars plana vitrectomy

INTERVENTIONS:
Procedure: Pars plana vitrectomy — All operations are performed in a similar fashion using the vitrectomy system with 23-gauge and 25-gauge vitrectomy probes. Surgical approach and technique include the use of tissue-staining dyes, choice of endotamponade, and postoperative face-down positioning regimen.
  Other Names: PPV

SUMMARY:
The goal of this clinical trial is to evaluate the visual and anatomical outcomes of large (410-1000 μm) full-thickness macular holes repair surgery using perfluoropropane (15% C3F8), sulfur hexafluoride (20% SF6) gas tamponade.

DETAILED DESCRIPTION:
The project is a randomized clinical trial with a follow up time of 6 months comparing the effects of surgical treatment of large (410-1000 μm) idiopathic macular holes. Patients are randomized to vitrectomy surgery with internal limiting membrane peeling using perfluoropropane (15% C3F8), sulfur hexafluoride (20% SF6) gas tamponad. Intra- and postoperative complications are registered.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 50 or above.
* Duration of Symptoms ≤ 12 months.
* Macular holes having a diameter 410-1000 μm.
* Informed consent.

Exclusion Criteria:

* Patients under 50 years of age.
* A patient who has already undergone treatment (surgery, laser etc.) for any disease of the retina.
* Traumatic or pediatric macular holes, and associated retinal detachment.
* History of any retinal disease such as high myopia, retinal dystrophies, central serous retinopathy, retinal vascular diseases, diabetic retinopathy, uveitis etc.
* Previous history of glaucoma or ocular hypertension.
* Failure to give informed consent.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Closure of macular holes | 6 months
  Closure of macular hole evaluated on optical coherence tomography
Type of macular hole closure | 6 months
  U-, V-, W-types of macular hole closure

SECONDARY OUTCOMES:
Best-corrected visual acuity | 6 months
  Visual acuity measured at last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- The Filatov Institute of Eye Diseases and Tissue Therapy, Odesa, Ukraine

IPD SHARING:
Plan to Share IPD: No